CLINICAL TRIAL: NCT00171067
Title: A Study to Evaluate the Effectiveness of Valsartan 320 mg in Combination With Lisinopril 20 mg Versus Monotherapy With Lisinopril 40 mg or Valsartan 320 mg in Hypertensive Patients With Microalbuminuria on the Reduction of Urinary Albumin Creatinine Ratio
Brief Title: VALERIA: Valsartan in Combination With Lisinopril in Hypertensive Patients With Microalbuminuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489ADE20
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Microalbuminuria, urinary albumin excretion, urinary albumin creatinine ratio, hypertension, valsartan, lisinopril, combination
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Lisinopril

INTERVENTIONS:
Drug: valsartan
Drug: lisinopril

SUMMARY:
The purpose of this study is to compare if the combination of valsartan 320 mg/lisinopril 20 mg versus the monotherapies of lisinopril 40 mg or valsartan 320 mg will result in a greater decrease of urinary albumin excretion measured as urinary albumin/creatinine ratio (UACR) in the first morning urine of hypertensive subjects with previously diagnosed microalbuminuria (MAU).

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate hypertension with a mean sitting diastolic blood pressure (MSDBP) > 85 and < 110 mmHg for non-treated patients. Previously treated patients with MSDBP < 110 mmHg. Treated is defined as having taken medication until < 2 days prior to Visit 1
* Positive urine spot test with Micral dipstick (detection of urinary albumin concentration of at least 50 mg/l) at Visit 1 (day -21).
* Confirmation of MAU of at least 2 out of 3 measurements determined in the first morning urine samples performed at Visit 1 day-21), Visit 2 (day -14) or Visit 3 (day -7). MAU is defined for male patients as urinary albumin creatinine ratio (UACR) > 2.5 mg/mmol and < 25.0 mg/mmol and for female patients as UACR > 3.5 mg/mmol and < 35.0 mg/mmol at both visits.

Exclusion Criteria:

* Evidence of renal impairment as determined by any one of the following:

  * serum creatinine clearance < 30 ml/min as determined by Cockroft and Gault formula [Cockroft and Gault, 1976] and/or
  * serum creatinine > 1.25 x ULN at Visit 1,
  * a history of dialysis, or
  * a history of nephrotic syndrome.
* Serum potassium values <3.5 mmol/l or >5.5 mmol/l at Visit 1
* Any medical condition which might significantly alter the urinary excretion of albumin

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary albumin excretion after 30 weeks

SECONDARY OUTCOMES:
Change from baseline in blood test for kidney function after 30 weeks
Reduction of urine albumin excretion in patients achieving blood pressures less than or equal to 130/80 mmHg
Change from baseline in circulating marker of inflammation after 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Investigative Centers, Germany
- Novartis Pharmaceuticals, Basel, Switzerland

REFERENCES:
- [Derived] Cooper TE, Teng C, Tunnicliffe DJ, Cashmore BA, Strippoli GF. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers for adults with early (stage 1 to 3) non-diabetic chronic kidney disease. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD007751. doi: 10.1002/14651858.CD007751.pub3. PMID 37466151
- [Derived] Menne J, Farsang C, Deak L, Klebs S, Meier M, Handrock R, Sieder C, Haller H. Valsartan in combination with lisinopril versus the respective high dose monotherapies in hypertensive patients with microalbuminuria: the VALERIA trial. J Hypertens. 2008 Sep;26(9):1860-7. doi: 10.1097/HJH.0b013e32830508aa. PMID 18698222